CLINICAL TRIAL: NCT03993223
Title: Scapular Kinematic and Shoulder Muscle Activity Alterations in Overhead Athletes With/Without Upper Trapezius Myofascial Trigger Point After Muscle Fatigue
Brief Title: Upper Trapezius Myofascial Trigger Point in Overhead Athletes After Upper Trapezius Muscle Fatigue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201904021RIND
Record Dates: First submitted 2019-06-12; First posted 2019-06-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Myofascial Trigger Point Pain; Fatigue
Keywords: Upper trapezius; Myofascial Trigger Point; Muscle fatigue; Overhead athlete
MeSH Terms: conditions — Myofascial Pain Syndromes; Fatigue

STUDY DESIGN:
Intervention Model Description: The treatment allocation and procedures involved in this randomized study were explained to all participants when they met inclusion criteria of VAS score of 4 or greater on the postoperative first day.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Data were collected by the attending surgeon who was blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTrP group (Experimental): Healthy overhead athletes with upper trapezius myofascial trigger point
  Interventions: Behavioral: Upper trapezius muscle fatigue
- Control group (Sham Comparator): Healthy overhead athletes without upper trapezius myofascial trigger point
  Interventions: Behavioral: Upper trapezius muscle fatigue

INTERVENTIONS:
Behavioral: Upper trapezius muscle fatigue — Isometric contraction of scapular elevation

SUMMARY:
The healthy overhead athletes with and without upper trapezius myofascial trigger point will be asked to perform a scapular elevation task until the upper trapezius muscle fatigue. The first hypothesis is that the subjects with upper trapezius myofascial trigger point will show significant difference in scapular kinematics and muscles activities when compared to subjects without upper trapezius myofascial trigger point. Besides, the investigators suggest that subjects with/without upper trapezius myofascial trigger point will show significant difference in scapular kinematics and muscles activities after upper trapezius muscle fatigue, especially in subjects with upper trapezius myofascial trigger point.

DETAILED DESCRIPTION:
The investigators will recruit healthy overhead athletes with and without upper trapezius myofascial trigger point. Participants will be asked to perform a sustained scapular elevation task at their peak force until the force decrease 50 %, which indicates upper trapezius muscle fatigue. There are two purposes in the current study: (1) to compare the differences between overhead athletes with/without upper trapezius myofascial trigger point during arm elevation in scapular kinematics and muscles activities (2) to investigate the effects of upper trapezius muscle fatigue on scapular kinematics and muscles activities in overhead athletes with/without upper trapezius myofascial trigger point. The first hypothesis is that the subjects with upper trapezius myofascial trigger point will show significant difference in scapular kinematics and muscles activities when compared to subjects without upper trapezius myofascial trigger point. Besides, the investigators suggest that subjects with/without upper trapezius myofascial trigger point will show significant difference in scapular kinematics and muscles activities after upper trapezius muscle fatigue, especially in subjects with upper trapezius myofascial trigger point. The outcome measurements includes scapular kinematics (upward/downward rotation, external/internal rotation, posterior/anterior tilting) and muscles activities (upper trapezius, serratus anterior, lower trapezius).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old active overhead athletes
* No symptoms in the shoulder of dominant side in the past 6 months
* Regularly perform overhead sports activity ≥ 3 hr/wk for more than 6 months

Exclusion Criteria:

* History of major shoulder/cervical injury or surgery in the past 6 months
* Experiencing shoulder pain, or participating in rehabilitation for shoulder pain in the past 6 months before the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Scapular kinematics | 10 minutes
  Change of scapular kinematics immediately after fatigue task
Scapular muscles electromyography | 10 minutes
  Change of scapular muscles electromyography immediately after fatigue task

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan university hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided